CLINICAL TRIAL: NCT05965869
Title: Creating Healthy Communities Through a Church-based, Community Health Worker-led Initiative
Brief Title: Healthy Communities Through CHW Initiatives
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Baylor College of Medicine (Other); University of Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0169; 23-0169 (Other: University of Texas Medical Branch, Galveston IRB)
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes program and education (Experimental): Receive diabetes program and education
  Interventions: Other: diabetes program

INTERVENTIONS:
Other: diabetes program — CHWs will contact participants weekly via phone or text, send bimonthly diabetes education videos, and provide optional monthly seminars.

SUMMARY:
Latino(a)s suffer from poor social determinants of health (SODH) conditions more than non-minority populations, and being a minority is risk factor alone for diabetes. In the proposed study, investigators will assist church members in becoming Community Health Workers (CHWs), train them in diabetes, and to track the ability to address healthcare access and quality barriers using an online platform.

DETAILED DESCRIPTION:
Social determinants of health (SODH) are environmental variables that determine quality-of-life outcomes and risks that are delineated into five domains. Inequities in SODH are directly associated with diabetes. Latino(a)s suffer from poor SODH conditions more than non-minority populations, and being a minority is risk factor alone for diabetes. To quantify progress in SODH, Healthy People 2030 has provided specific objectives to measure each domain (economic stability, education access and quality, healthcare access and quality, neighborhood and build environment, and social and community context); this application focuses on the healthcare access and quality domain. While there are numerous screening mechanisms to identify SODH conditions, there is a critical need to implement interventions that are translatable into real-world practices.

A successful intervention requires several components. For the community, sites are needed that can bring individuals together, making collaboration with faith-based establishments of particular interest. Religious institutions provide an infrastructure that will persist beyond funding periods and a framework for the community to share a responsibility of health promotion. Churches also provide an accessible and familiar setting to provide health outreach programs but often lack trained personnel to conduct initiatives. In addition, training leaders within these settings who can reach the community is essential. Community Health Workers (CHWs) are trusted leaders within their community. Training church members to become CHWs potentially establishes a site familiar to the surrounding communities led by trusted individuals who understand the population at hand. Finally, secure avenues to collect and transmit data are needed. Utilizing secure HIPAA-approved technology reduces risks of loss of confidentiality while allowing collection of valuable information that may not have been collected otherwise. Since COVID-19, investigators have increased the use of online platforms, but these modalities must be translatable to personnel with potentially little to no technological experience.

To address gaps in SDOH, the investigators propose a 6-month church-based intervention for Latino(a)s with and at risk for diabetes (n=460) in a two phase study, pilot followed by main study. We will assist church members in becoming CHWs, train them in diabetes, and use an online platform to track the ability to address healthcare access and quality barriers. The research team will provide telementoring to local community teams (church leadership and CHWs) to initiate the intervention. We will test the feasibility of the program using three pre-established areas of focus: acceptability, integration, limited efficacy testing.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking Latino(a)s adults

Exclusion Criteria:

* pregnant state or anticipated state in the next 6 months
* Type 1 diabetes diagnosis
* Not geographically located to reach church site/attend classes
* Not Spanish-speaking, and
* Self-disclosed diagnosis of schizophrenia, psychotic/delusional disorder, or severe Alzheimer's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the integration of the intervention | 6-months
  CHW ability to use software as measured by the number of anticipated vs. actual documents uploaded at 6-months

SECONDARY OUTCOMES:
Provide acceptability data of the intervention | 6-months
  Site, CHW, and participant survey data at 6-months as measured on a Likert scale, e.g., Likert scale from 1 to 5 where 1 is unsatisfied and 5 is very satisfied.
  Participant participation trends in the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Vaughan, DO, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wyatt LC, Katigbak C, Riley L, Zanowiak JM, Ursua R, Kwon SC, Trinh-Shevrin C, Islam NS. Promoting Physical Activity Among Immigrant Asian Americans: Results from Four Community Health Worker Studies. J Immigr Minor Health. 2023 Apr;25(2):291-305. doi: 10.1007/s10903-022-01411-y. Epub 2022 Oct 23. PMID 36273386
- [Background] Hessler D, Fisher L, Dickinson M, Dickinson P, Parra J, Potter MB. The impact of enhancing self-management support for diabetes in Community Health Centers through patient engagement and relationship building: a primary care pragmatic cluster-randomized trial. Transl Behav Med. 2022 Oct 7;12(9):909-918. doi: 10.1093/tbm/ibac046. PMID 36205473
- [Background] Levy NK, Park A, Solis D, Hu L, Langford AT, Wang B, Rogers ES. Social Determinants of Health and Diabetes-Related Distress in Patients With Insulin-Dependent Type 2 Diabetes: Cross-sectional, Mixed Methods Approach. JMIR Form Res. 2022 Oct 12;6(10):e40164. doi: 10.2196/40164. PMID 36222807
- [Background] Wagner J, Bermudez-Millan A, Buckley T, Buxton OM, Feinn R, Kong S, Kuoch T, Nye LM, Scully M. Self-reported outcomes of a randomized trial comparing three community health worker interventions for diabetes prevention among Cambodian Americans with depression. Patient Educ Couns. 2022 Dec;105(12):3501-3508. doi: 10.1016/j.pec.2022.09.011. Epub 2022 Oct 6. PMID 36307274
- [Background] Deverts DJ, Heisler M, Kieffer EC, Piatt GA, Valbuena F, Yabes JG, Guajardo C, Ilarraza-Montalvo D, Palmisano G, Koerbel G, Rosland AM. Comparing the effectiveness of Family Support for Health Action (FAM-ACT) with traditional community health worker-led interventions to improve adult diabetes management and outcomes: study protocol for a randomized controlled trial. Trials. 2022 Oct 3;23(1):841. doi: 10.1186/s13063-022-06764-1. PMID 36192769
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Keegan CN, Johnston CA, Cardenas VJ Jr, Vaughan EM. Evaluating the Impact of Telehealth-Based, Diabetes Medication Training for Community Health Workers on Glycemic Control. J Pers Med. 2020 Sep 11;10(3):121. doi: 10.3390/jpm10030121. PMID 32932865
- [Background] Garcia AA, Villagomez ET, Brown SA, Kouzekanani K, Hanis CL. The Starr County Diabetes Education Study: development of the Spanish-language diabetes knowledge questionnaire. Diabetes Care. 2001 Jan;24(1):16-21. doi: 10.2337/diacare.24.1.16. PMID 11194219
- [Background] Dumville JC, Torgerson DJ, Hewitt CE. Reporting attrition in randomised controlled trials. BMJ. 2006 Apr 22;332(7547):969-71. doi: 10.1136/bmj.332.7547.969. PMID 16627519
- [Background] Parmanto B, Lewis AN Jr, Graham KM, Bertolet MH. Development of the Telehealth Usability Questionnaire (TUQ). Int J Telerehabil. 2016 Jul 1;8(1):3-10. doi: 10.5195/ijt.2016.6196. eCollection 2016 Spring. PMID 27563386
- [Background] Belone L, Lucero JE, Duran B, Tafoya G, Baker EA, Chan D, Chang C, Greene-Moton E, Kelley MA, Wallerstein N. Community-Based Participatory Research Conceptual Model: Community Partner Consultation and Face Validity. Qual Health Res. 2016 Jan;26(1):117-35. doi: 10.1177/1049732314557084. Epub 2014 Oct 31. PMID 25361792
- [Background] Rimawi A, Shah A, Louis H, Scales D, Kheiran JA, Jawabreh N, Yunez S, Horino M, Seita A, Wispelwey B. Community Health Worker Program Outcomes for Diabetes and Hypertension Control in West Bank Refugee Camps: A Retrospective Matched Cohort Study. Glob Health Sci Pract. 2022 Oct 31;10(5):e2200168. doi: 10.9745/GHSP-D-22-00168. Print 2022 Oct 31. PMID 36316145
- [Background] Vaughan EM, Johnson E, Naik AD, Amspoker AB, Balasubramanyam A, Virani SS, Ballantyne CM, Johnston CA, Foreyt JP. Long-Term Effectiveness of the TIME Intervention to Improve Diabetes Outcomes in Low-Income Settings: a 2-Year Follow-Up. J Gen Intern Med. 2022 Sep;37(12):3062-3069. doi: 10.1007/s11606-021-07363-7. Epub 2022 Feb 7. PMID 35132555
- [Background] Vaughan EM, Naik AD, Amspoker AB, Johnston CA, Landrum JD, Balasubramanyam A, Virani SS, Ballantyne CM, Foreyt JP. Mentored implementation to initiate a diabetes program in an underserved community: a pilot study. BMJ Open Diabetes Res Care. 2021 Aug;9(1):e002320. doi: 10.1136/bmjdrc-2021-002320. PMID 34385148

DOCUMENTS (1):
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT05965869/ICF_000.pdf